CLINICAL TRIAL: NCT06140043
Title: Augmented Reality for Orthognatic Surgery Patient Education
Acronym: NARRATE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: UMC Utrecht (Other); Uniklinik RTWH Aachen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17618
Record Dates: First submitted 2023-10-25; First posted 2023-11-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Malocclusion; Dentofacial Deformities; Patient Satisfaction; Informed Consent; Patient Education
Keywords: Orthognatic Surgery; Augmented Reality; Patient Satisfaction; Informed Consent; Patient Education; 3D; BSSO; BIMAX
MeSH Terms: conditions — Malocclusion; Dentofacial Deformities; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: patients are randomised to one of two groups, either consultation with models on a computer screen or with models shown in augmented reality
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitor (Active Comparator): Patient consultation with 3D models of bone and skin, seen with a monitor screen
  Interventions: Other: Patient consultation
- Augmented Reality (Experimental): Patient consultation with 3D models of bone and skin, seen in augmented reality trough AR glasses
  Interventions: Other: Patient consultation

INTERVENTIONS:
Other: Patient consultation — Providing information about the current clinical problem of orthognatic surgery patients and the proposed treatment for it.

SUMMARY:
To evaluate whether the use of augmented reality (AR) for visualizing 3D models can be a valuable addition to patient education regarding orthognathic procedures compared to using only 2D visualization (on a computer screen).

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for an orthognathic intake consult in the period of July to april 2024 at the UMCU or UMCG or Uniklinik RTWH Aachen;
* Patients with dentofacial deformity (dysgnathia) including: class II malocclusion, class III malocclusion, or open bite;
* Patients undergoing treatment using BSSO (Bilateral Sagittal Split Osteotomy), Le Fort I, or BIMAX;
* The planned treatment is either with or without a genioplasty procedures.
* Patients 16 years of age or older.

Exclusion Criteria:

* Patients with craniofacial syndromes, such as cleft lip and palate
* Patient which require an osteotomy involving two or more segments

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Immediately after the regular first intake consult
  Patient satisfaction of the intake consult. Focussed on the explanation of the condition and proposed treatment, measured through a questionnaire. The questionnaire measures the clarity and importance of the information for the patient. For both parameters a median score will be calculated between 0 and 5
Objective knowledge | Immediately after the regular first intake consult
  Patient knowledge of the medical problem and proposed treatment, also measured by a questionnaire. Patient can get 2 points when all four question are right, if all questions are answered incorrectly, then -2 points

OTHER OUTCOMES:
Diagnosis | During the first intake consult
  Orthognatic diagnosis
Occlusion Class | During the first intake consult
  Class of the occlusion of the patient before surgery

CONTACTS AND LOCATIONS:
Overall Officials: J Kraeima, dr., Principal Investigator — UMC Groningen
Locations (3):
- UniKlinik RWTH Aachen, Aachen, Germany
- Netherlands (2):
  - UMC Groningen, Groningen, Provincie Groningen
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No